CLINICAL TRIAL: NCT05958784
Title: A Pilot Study for the PKU Carriers Trial: Evaluating the Impact of PKU Carrier Status on Cognition, Mental Health, Blood Pressure and L-phenylalanine Metabolism
Brief Title: PKU Carriers Trial (Pilot Study): Impact on Cognition, Mental Health, Blood Pressure and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Justine Keathley, Assistant Professor, University of Guelph
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REB23-03-017
Record Dates: First submitted 2023-07-05; First posted 2023-07-25 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Autosomal Recessive Disorder (Genetic Carriers of PKU)
MeSH Terms: interventions — Phenylalanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Genetic Carriers and Non-Carriers of PKU (Experimental)
  Interventions: Dietary Supplement: L-Phenylalanine

INTERVENTIONS:
Dietary Supplement: L-Phenylalanine — 100 mg/kg

SUMMARY:
This is a clinical intervention pilot/feasibility study of PKU carriers (cases) and non-carriers (controls). Upon completing the informed consent process, participants will complete baseline measures of chronic mental health prior to the intervention (PHQ-9, GAD-7, BIS-Brief). Participants will attend the Human Nutraceutical Research Unit (HNRU) at the University of Guelph, fasted, and first undergo baseline measures of cognition and acute mental health (mood) and provide samples or saliva, urine and dried blood spots to evaluate phenylalanine (Phe), tyrosine (Tyr) and their metabolites (PAH pathway functioning). Participants will also complete a brief questionnaire which will include age, sex, ethnicity, income, weight and height (measured using a stadiometer and calibrated weigh scale), and confirmation that participants arrived to the lab fasted (i.e. have only had water to drink and no other foods/beverages prior to analyses). Blood pressure will also be measured at baseline. Following baseline tests, participants will consume a pure L-Phe supplement dosed at 100 mg/kg mixed into 250 mL water with 1 tsp white sugar. Blood pressure will be repeated at 1-hour post-L-Phe consumption. Two-hours postprandial, participants will repeat the cognitive tests and acute mental health (mood) assessment, blood pressure measurement and provide follow-up saliva, urine and dried blood spot samples. Participants will also be asked to report any side effects they experienced with the L-Phe consumption.

ELIGIBILITY:
Inclusion Criteria:

* Known carrier or non-carrier of PKU
* At least 18 years of age
* Comfortable fasting the morning of the study (no food or drink other than water)

Exclusion Criteria:

* Diagnosed with: PKU, severe neurodegenerative conditions affecting cognition (e.g. Alzheimer's, Parkinson's, dementia), melanoma, hypertension, liver disease and/or kidney disease
* Taking a Monoamine Oxidase Inhibitor anti-depressant
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Stop Signal Reaction Time (Response Inhibition) | Change from baseline to 2-hours post L-Phe supplementation

SECONDARY OUTCOMES:
Working Memory | Change from baseline to 2-hours post L-Phe supplementation
  N-Back Test Outcome
Stop Signal Delay | Change from baseline to 2-hours post L-Phe supplementation
  Stop Signal Task Outcome
Individual Coefficient of Variance (Variability in Reaction Times) | Change from baseline to 2-hours post L-Phe supplementation
  Stop Signal Task Outcome
Phenylalanine Levels | Change from baseline to 2-hours post L-Phe supplementation
Tyrosine Levels | Change from baseline to 2-hours post L-Phe supplementation
Phenylalanine Metabolites: e.g.phenylethylamine, tyramine, phenylpyruvate, others | Change from baseline to 2-hours post L-Phe supplementation
Tyrosine Metabolites: e.g. L-DOPA, dopamine, norepinephrine, epinephrine, p-hydroxyphenylpyruvate, homogentisic acid, fumarate, others | Change from baseline to 2-hours post L-Phe supplementation
Mood | Change from baseline to 2-hours post L-Phe supplementation
  Profile of Mood States (POMS) Outcome
Blood Pressure | Change from baseline to 1-hour and 2-hours post L-Phe supplementation
  Systolic and Diastolic

OTHER OUTCOMES:
Chronic Anxiety | Baseline
  GAD-7 Outcome
Chronic Depression | Baseline
  PHQ-9 Outcome
Impulsivity | Baseline
  BIS-Brief Outcome
Trial-by-trial analysis | Change from baseline to 2-hours post L-Phe supplementation
  To be conducted if there are significant findings from the four main stop signal task outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No